CLINICAL TRIAL: NCT01484873
Title: Effects of Exenatide on Body Weight in Patients With Hypothalamic Obesity
Brief Title: Weight Loss Study for Patients With Obesity Due to Craniopharyngioma or Other Brain Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ashley Shoemaker, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111185
Record Dates: First submitted 2011-10-20; First posted 2011-12-02 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Obesity; Overweight; Craniopharyngioma
Keywords: Exenatide; Byetta; Hypothalamic Obesity; Obesity; Craniopharyngioma
MeSH Terms: conditions — Obesity; Overweight; Craniopharyngioma; Sexual Infantilism | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exenatide (Experimental): All patients received exenatide 10mcg BID x 50 weeks
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Treatment with exenatide 5 mcg twice daily for 4 weeks, then 10 mcg twice daily for 46 weeks.
  Other Names: Byetta

SUMMARY:
The purpose of this study is to determine whether exenatide can cause weight loss in patients with a history of craniopharyngioma or other brain lesion.

DETAILED DESCRIPTION:
Hypothalamic obesity occurs in up to 60% of patients with tumors in the hypothalamic region, most commonly craniopharyngiomas. Hypothalamic dysfunction can be due to tumor infiltration and as a consequence of surgery or radiation therapy. Survivors who develop obesity have greater morbidity and mortality than normal weight survivors. Prevention and treatment of obesity in this population is vital in order to decrease the morbidity and mortality from diabetes, stroke and myocardial infarction.

Exenatide (Byetta®) is a GLP-1 homologue that was FDA approved for treatment of type 2 diabetes in 2005. It also decreases the rate of gastric emptying and increases satiety and has been shown to cause weight loss in some people. Exenatide may improve insulin sensitivity and satiety in patients with hypothalamic obesity but without the risks of bariatric surgery. The investigators hypothesize that treatment with exenatide will lead to weight loss in patients with hypothalamic obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years old
* History of craniopharyngioma or other lesion in the hypothalamic region
* Greater than 6 months post-treatment, including chemotherapy, surgery or radiation
* BMI >30 mg/m2
* Females must be post-menopausal, surgically sterile or using effective birth control for at least 12 weeks

Exclusion Criteria:

* HgbA1C >7%
* Use of diabetes medications other than metformin in the past 12 weeks, including exenatide
* Use of weight loss drugs or initiation of a weight loss program in past 3 months
* Impaired renal function or history of kidney transplant
* History of gall stones (unless s/p cholecystectomy), pancreatitis or alcoholism
* Personal or family history of medullary carcinoma of the thyroid or MEN type 2
* History of gastroparesis or other gastric motility problems as exenatide decreases gastric motility
* History of allergic reaction to exenatide or other medication components
* Other significant comorbidities other than pituitary deficiencies
* Currently prescribed warfarin (exenatide may alter warfarin metabolism)
* Pregnant or lactating females
* History of severe hypoglycemia (BG <60 and requiring assistance from another person)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Shoemaker, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lomenick JP, Buchowski MS, Shoemaker AH. A 52-week pilot study of the effects of exenatide on body weight in patients with hypothalamic obesity. Obesity (Silver Spring). 2016 Jun;24(6):1222-5. doi: 10.1002/oby.21493. Epub 2016 May 2. PMID 27133664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University clinics and online advertisements from June, 2012 - March, 2013
Groups:
- Exenatide: exenatide 10 mcg twice daily
Period: Overall Study
Arm/Group | Exenatide
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Exenatide
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 8
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Weight [Mean (Standard Deviation); unit: kg] | 137.2 (37.6)
Resting energy expenditure [Mean (Standard Deviation); unit: kcal/day] | 2215.0 (654.9)
Satiety [Mean (Standard Deviation); unit: mm] — minimum 0, maximum 100
  mm | 68.9 (15.4)
Insulin AUC [Mean (Standard Deviation); unit: 120 min*uU/mL] | 13076 (7482)
Gastric emptying half life [Mean (Standard Deviation); unit: minutes] | 175.4 (81.0)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight (kg)
Description: Change in body weight from baseline to end of study
Time Frame: baseline, 50 weeks
Population: Patients that completed the study
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Exenatide
Number analyzed (Participants) | 8
kg | -1.4 [-2.2 to 4.9]

2. Secondary Outcome: Resting Energy Expenditure (Kcals Per Day)
Description: Change in resting energy expenditure from baseline to 50 weeks
Time Frame: baseline, 50 weeks
Population: 8 patients completed the study but one patient did not have REE data available due to technical difficulties
Measure: Mean (95% Confidence Interval); unit: kcal/day
Arm/Group | Exenatide
Number analyzed (Participants) | 7
kcal/day | -157.7 [-766.1 to 450.6]

3. Secondary Outcome: Visual Analogue Scales for Post-meal Satiety
Description: Change in visual analogue scales scores from baseline to 50 weeks. Higher score indicates greater satiety (minimum 0, maximum 100).
Time Frame: baseline, 50 weeks
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Exenatide
Number analyzed (Participants) | 8
mm | -2.5 [-19.7 to 14.7]

4. Secondary Outcome: Insulin Secretion (Area Under the Curve)
Description: Change in insulin secretion from baseline
Time Frame: baseline, 50 weeks
Measure: Mean (95% Confidence Interval); unit: 120 min*uU/mL x
Arm/Group | Exenatide
Number analyzed (Participants) | 8
120 min*uU/mL x | -89.3 [-5127 to 4948]

5. Secondary Outcome: Gastric Emptying Rate (13C-octanoic Acid Isotope Excretion Half Life)
Description: Change in the isotope excretion half life during a gastric emptying test at baseline and at 50 weeks
Time Frame: baseline, 50 weeks
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Exenatide
Number analyzed (Participants) | 8
minutes | 12.9 [-38.5 to 64.3]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Exenatide
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=10)
Nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hypoglycemia (Endocrine disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 3 (3)
Irregular heart beat (Cardiac disorders) | 1 (1)
Acute otitis media (Ear and labyrinth disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
kidney stones (Renal and urinary disorders) | 1 (1)
URI (Infections and infestations) | 3 (4)
Nose bleed (Blood and lymphatic system disorders) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 2 (2)
strep throat (Infections and infestations) | 1 (1)
tingling/numbness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes